CLINICAL TRIAL: NCT02806830
Title: Evaluation de la gêne Oculaire après Injections intravitréennes
Brief Title: Ocular Discomfort Assessment After Intravitreal Injections
Acronym: EVAGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Oudy SEMOUN, Doctor in ophtalmology, Centre Hospitalier Intercommunal Creteil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EVAGO
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Macular Degeneration; Diabetic Retinopathy; Retinal Artery Occlusion; Myopia, Degenerative
Keywords: Intravitreal injection; AMD; Diabetic Retinopathy; Retinal Artery Occlusion; Myopia, Degenerative; eye drops
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy; Retinal Artery Occlusion; Myopia, Degenerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optive after the second anti-VEGF injection (Experimental): Naive patients requiring intravitreal injection. Patients will be enrolled in this study within the 2 first intravitreal injections to assess quality of life and ocular discomfort without wetting agent (ie after the first injection) and with wetting agent (ie after the second injection)
  Interventions: Drug: Optive

INTERVENTIONS:
Drug: Optive — Optive eye drops will be prescribed to each included patients after their second intravitreal injection; patients will received 1 drop in the affected eye 2 times a day during 3 days

SUMMARY:
In this study, ocular discomfort following intravitreal injection in naïve patients will be studied, as well as the efficacy of wetting agent (Optive eyewash) to prevent ocular discomfort.

DETAILED DESCRIPTION:
In naive patients, the two first intravitreal injections will be studied. Within the first injection, no wetting agent will be delivered. Within 72hours after this first intravitreal injections, patients will be contacted by phone by a nurse to complete questionnaires on quality of life and on ocular pain and eye discomfort.

After the second injection, a treatment with wetting agent will be prescribed. With 72hours after the second injection, quality of life, ocular discomfort as well as acceptability and tolerance of the eye drops will also be assessed by a phone questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with social healthcare
* Patient understanding French language
* Patient requiring anti-VEGF treatment by intravitreal injection

Exclusion Criteria:

* Patient treated by Ozurdex® before
* Patient with known and treated ocular dryness
* Non naive patient for intravitreal injection
* Hypersensitivity to Carmellose
* Patient who received wetting agent within the 3 last months
* History of povidone-iodine allergy
* Pregnant or breastfeeding mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the overall scores of the ocular discomfort questionnaire after the 2 first intravitreal injection in naïve patients | within the 72h after the first and the second intravitreal injections

CONTACTS AND LOCATIONS:
Overall Officials: Oudy SEMOUN, MD, Principal Investigator — CHI Créteil
Locations (1):
- Chi Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ba J, Peng RS, Xu D, Li YH, Shi H, Wang Q, Yu J. Intravitreal anti-VEGF injections for treating wet age-related macular degeneration: a systematic review and meta-analysis. Drug Des Devel Ther. 2015 Sep 28;9:5397-405. doi: 10.2147/DDDT.S86269. eCollection 2015. PMID 26451092
- [Background] Pe'er J, Folberg R, Itin A, Gnessin H, Hemo I, Keshet E. Vascular endothelial growth factor upregulation in human central retinal vein occlusion. Ophthalmology. 1998 Mar;105(3):412-6. doi: 10.1016/S0161-6420(98)93020-2. PMID 9499769
- [Background] Nghiem-Buffet S, Cohen SY. [Retinal vein occlusion: anti-VEGF treatments]. J Fr Ophtalmol. 2009 Nov;32(9):679-86. doi: 10.1016/j.jfo.2009.10.002. Epub 2009 Oct 29. French. PMID 19879018
- [Background] Salam A, DaCosta J, Sivaprasad S. Anti-vascular endothelial growth factor agents for diabetic maculopathy. Br J Ophthalmol. 2010 Jul;94(7):821-6. doi: 10.1136/bjo.2009.163576. Epub 2009 Jun 24. PMID 19556214
- [Background] Massin P, Bandello F, Garweg JG, Hansen LL, Harding SP, Larsen M, Mitchell P, Sharp D, Wolf-Schnurrbusch UE, Gekkieva M, Weichselberger A, Wolf S. Safety and efficacy of ranibizumab in diabetic macular edema (RESOLVE Study): a 12-month, randomized, controlled, double-masked, multicenter phase II study. Diabetes Care. 2010 Nov;33(11):2399-405. doi: 10.2337/dc10-0493. PMID 20980427
- [Background] Stewart MW. The clinical utility of aflibercept for diabetic macular edema. Diabetes Metab Syndr Obes. 2015 Sep 18;8:473-82. doi: 10.2147/DMSO.S72792. eCollection 2015. PMID 26425104
- [Background] Massamba N, Elluard M, Agoune W, Guyader V, Ingram A, Pasquier B, Knoeri J. Assessment of ocular pain following ranibizumab intravitreal injection. Acta Ophthalmol. 2015 May;93(3):e231-2. doi: 10.1111/aos.12531. Epub 2014 Aug 13. No abstract available. PMID 25123226
- [Background] Meyer CH, Krohne TU, Charbel Issa P, Liu Z, Holz FG. Routes for Drug Delivery to the Eye and Retina: Intravitreal Injections. Dev Ophthalmol. 2016;55:63-70. doi: 10.1159/000431143. Epub 2015 Oct 26. PMID 26501462